CLINICAL TRIAL: NCT02212613
Title: Protocol 331-13-004: An Exploratory, Multicenter, Single-blind, fMRI Study of Fixed-dose Brexpiprazole (OPC 34712) (2 mg/Day Tablets) as an Adjunctive Treatment
Brief Title: Brexpiprazole (OPC 34712) Trial in the Treatment of Adults With Major Depressive Disorder and Irritability
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 331-13-004
Record Dates: First submitted 2014-07-23; First posted 2014-08-08 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Major Depressive Disorder and Irritability
Keywords: Major Depressive Disorder; Mental Disorders, nonpsychotic episode, antipsychotic; Mood Disorder, psychotic disorder
MeSH Terms: conditions — Depressive Disorder, Major; Mental Disorders; Affective Disorders, Psychotic | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole (Experimental): Brexpiprazole - Up to 2 mg/day, once daily dose, tablets, orally
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Treatment (6 weeks) Up to 2 mg/day, once daily dose, tablets, orally
  Other Names: OPC-34712

SUMMARY:
The purpose of this study is to explore the effects of fixed-dosed brexpiprazole adjunctive treatment in subjects with Major Depressive Disorder with irritability

ELIGIBILITY:
* Inclusion Criteria:

  * Are 18 to 55 years of age, inclusive, at the time of informed consent with a diagnosis of a single or recurrent, nonpsychotic episode of MDD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR™) and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.) and an adequate clinical psychiatric evaluation
  * Have received a single, trial-approved SSRI or SNRI at an adequate dose for ≥ 6 weeks prior to screening
  * Have a treatment history of inadequate ADT response to at least one ADT (but not > 3) for the current episode. The current major depressive episode must be ≥ 6 weeks in duration. (An inadequate ADT response is defined as < 50% reduction in depressive symptom severity, as measured by subject self-report on the MGH-ATRQ.)
  * To be eligible for this trial

    * Have a MADRS Total Score of 20 or more at screening and the Phase A baseline, and have a MADRS Total Score of 18 or more at the Phase B baseline
    * Have no more than 20% improvement in MADRS Total Score at Phase B baseline compared to Phase A baseline
    * Have a score of 6 or more on the KSQ based on the Well being and Reversal Distress Anger-hostility subscales at screening, Phase A baseline, and Phase B baseline
    * Have anger attacks as documented by the AAQ at screening, Phase A baseline, and Phase B baseline
  * Are right-handed (defined according to the Edinburgh Handedness Inventory) and have normal hearing and normal/corrected-to-normal vision
  * Are willing to discontinue all prohibited psychotropic medications to meet protocol-required washouts prior to and during the trial period
  * Eligibility confirmed through a telephone SAFER interview with the subject and an independent expert centralized rater
* Exclusion Criteria:

  * Have a current need for involuntary commitment or have been hospitalized within 4 weeks of screening for the current major depressive episode
  * Have a current DSM-IV-TR Axis I diagnosis of any of the following: delirium, dementia, amnestic, or other cognitive disorders; schizophrenia, schizoaffective disorder, or other psychotic disorders; bipolar I disorder, bipolar II disorder, or bipolar disorder not otherwise specified; eating disorders (including anorexia nervosa or bulimia); obsessive compulsive disorder; panic disorder; or post-traumatic stress disorder
  * Have any of the following current Axis II DSM-IV-TR diagnoses: borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorders, or mental retardation
  * Experiencing hallucinations, delusions, or any psychotic symptomatology in the current major depressive episode

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Phase B baseline to Phase B Week 6 in functional magnetic resonance imaging (fMRI) BOLD activation score in the ventromedial prefrontal cortex and amygdala, scanned by fMRI during performance of the Emotion-induction Task | Week 6

SECONDARY OUTCOMES:
Change from Phase B baseline to Phase B Week 6 in Montgomery Asberg Depression Rating Scale (MADRS) Total Score | Week 6
Change from Phase B baseline to Phase B Week 6 in Spielberger State Trait Anger Expression Inventory (STAXI-2) Part 1 | Week 6
Change from Phase B baseline to Phase B Week 6 in Visual Analog Scale (VAS) | Week 6
Change from Phase B baseline to Phase B Week 6 in Clinical Global Impression - Severity of Illness Scale (CGI-S) score | Week 6
Clinical Global Impression - Improvement Scale (CGI-I) score at Phase B Week 6 | Week 6
MADRS response rate, where response is defined as ≥ 50% reduction in respective total scores from Phase B baseline to Phase B Week 6 | Week 6
MADRS remission rate, where remission is defined as MADRS Total Score ≤ 10 and 50% reduction in MADRS Total Score from Phase B baseline to Phase B Week 6 | Week 6
Change from Phase B baseline to Phase B Week 6 in Sheehan Disability Scale (SDS) 3-item mean score | Week 6
Change from Phase B baseline to Phase B Week 6 in Anger Attacks Questionnaire (AAQ) score | Week 6
Change from Phase B baseline to Phase B Week 6 in Symptoms of Depression Questionnaire (SDQ) | Week 6
Change from Phase B baseline to Phase B Week 6 in Kellner Symptom Questionnaire (KSQ) | Week 6
Change from Phase B baseline to Phase B Week 6 in Barratt Impulsiveness Scale 11 item (BIS-11) Total Score | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd Japan (OPCJ)
Locations (1):
- Emory University, Atlanta, Georgia, United States